CLINICAL TRIAL: NCT06433440
Title: An Open-label, Randomized Study Evaluating the Safety and Immunogenicity of the Purified Vero Cell Rabies Vaccine PVRV Administered Intradermally and Intramuscularly as Post-exposure Prophylaxis
Brief Title: Safety and Immunogenicity of Purified Verocell Rabies Vaccine PVRV Administered Intramuscularly and Intradermally
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Peshawar (Other)
Collaborators: Hayatabad Medical Complex (Other Government)
Responsible Party: Principal Investigator, Mohammad Ismail, Dr. Mohammad Ismail Associate Professor of Clinical Pharmacy, University of Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PVRV-ID
Record Dates: First submitted 2024-05-13; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-1 (Experimental): 0.2 ml of PVRV Intradermally (ID) on the following days: Day0, Day3, and Day7
  Biological: PVRV
  PEP regimen
  Interventions: Biological: PVRV
- Group-2 (Experimental): 0.5 ml of PVRV Intramuscularly (IM) on the following days: Day0, Day3, and Day7, Day14 and Day28
  Biological: PVRV
  PEP regimen
  Interventions: Biological: PVRV

INTERVENTIONS:
Biological: PVRV — Group-1 will receive PVRV ID on on the following days: Day0, Day3, Day7, while group-2 will receive PVRV IM on Day0, Day3, Day7, Day14, and Day28.

SUMMARY:
Rabies is fatal disease but preventable with rabies vaccines and immunoglobulins, conventionally involves intramuscular (IM) administration of the vaccine. However, switching the intradermal (ID) route offers potential advantages in dosing, time and cost without compromising efficacy and safety. Therefore, this study aims to compare the safety and immunogenicity of a short-term three-doses intradermal regimen (3D-ID) with a conventional five-doses intramuscular regimen (5D-IM) of the purified Vero cell rabies vaccine (PVRV), administered via both intramuscular (IM) and intradermal (ID) routes as post-exposure prophylaxis (PEP).

DETAILED DESCRIPTION:
Rabies vaccines can be used ID for PEP, according to a WHO Expert Committee recommendation. The administration of short-term PEP through ID (3-doses) offers a safe, immunogenic, dose-sparing, and cost-effective alternative to the conventional protocol (IM, 5-dose regimen) while reducing the volume by up to 60 to 80% and vaccination schedules by 3 weeks. This strategy has the potential to reduce the overall requirement and cost of such vaccines, along with minimizing the burden on healthcare professionals and facilities. Furthermore, this strategy is more likely to improve vaccination compliance compared to conventional protocol, and will certainly improve treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 2 year or older
* Both male and female
* Dog-bite cases only
* Informed consent form signed by the individual participant and/or their parents or guardian in case of minor age or major Trauma

Exclusion Criteria:

* Subject is participating in any other clinical trial.
* Pregnant and lactating women
* Have a plan to donate blood while participating in the study
* Received any other vaccine except rabies vaccines in last 6 months

Ages: 2 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy of PVRV administered intradermally vs intramuscularly based on immune response. | 56 days
  Patients were assigned into two groups each consisting of n=50 patients: Group-1 and Group-2. Group-1 were administered PVRV intradermally in a dose of 0.2ml on day 0, day 3, and day 7 as post exposure prophylaxis. While, patients in the group-2 received PVRV intramuscularly in a dose of 0.5ml on day 0, day 3, day 7, day 14 and day 28.
  Efficacy of PVRV in both groups were measured by the presence of rabies virus neutralizing antibodies (RVNA). Patients with an RVNA titer of ≥ 0.5 IU/mL were considered immunized.

SECONDARY OUTCOMES:
To evaluate the safety of PVRV administered intradermally and intramuscularly based on the frequency of adverse drug events | 42 days
  Monitoring of both local and systemic adverse events occurring during the study period The safety of the PVRV was determined by reviewing ADEs obtained during physical examinations following vaccine administration and during follow-up visits in both the groups (group-1 and group-2). The ADEs were recorded after completion of the full vaccination schedule by following-up the patient until day 42. Adverse drug events were characterized in terms of local and systemic effects. A reaction was considered local when it occurred at the site of injection within a few hours of administration, while systemic effects were defined as those occurring in tissues distant from the site of contact between the body and vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ismail, PhD, Study Chair — Department of Pharmacy, University of Peshawar; Waqar Ali, MPhil, Study Director — Department of Pharmacy University of Peshawar
Locations (1):
- Mohammad Ismail, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
Will be shared on reasonable request from the PI